CLINICAL TRIAL: NCT04810520
Title: Live Stream of Prehospital point-of Care Ultrasound by Air Rescue Physicians
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled due to organizational problems
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Clinical Investigator, Medical University of Vienna
Other Study IDs: 1218/2021
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Echocardiography; Telemedicine
Keywords: Ultrasound diagnostics; Prehospital emergency medicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Point-of-care ultrasound with tele-supervision: Point-of-care ultrasound of critically ill patients (acute dyspnoea, circulatory failure, trauma) will be performed with tele-supervision.
  Interventions: Other: Point-of-care ultrasound with tele-supervision
- Point-of-care ultrasound without tele-supervision: Point-of-care ultrasound of critically ill patients (acute dyspnoea, circulatory failure, trauma) will be performed without tele-supervision.
  Interventions: Other: Point-of-care ultrasound without tele-supervision

INTERVENTIONS:
Other: Point-of-care ultrasound with tele-supervision — Point-of-care ultrasound of critically ill patients (acute dyspnoea, circulatory failure, trauma) will be performed with tele-supervision.
  Groups: Point-of-care ultrasound with tele-supervision
Other: Point-of-care ultrasound without tele-supervision — Point-of-care ultrasound of critically ill patients (acute dyspnoea, circulatory failure, trauma) will be performed with tele-supervision.
  Groups: Point-of-care ultrasound without tele-supervision

SUMMARY:
Background: Point-of-care ultrasound (POCUS) has been suggested as a useful tool in emergency medicine for diagnosis and treatment of reversible causes. However, in prehospital setting performing ultrasound and the translation of the findings can be challenging. As new prehospital ultrasound devices offer the possibility for remote supervision, the impact of tele-supervision on time to diagnosis of critically ill patients is unclear.

Aims: The aim of this study is to evaluate the impact of tele-supervision on the time of POCUS in prehospital critically ill patients by air rescue physicians.

Methods: In total 100 critically ill patients suffering from acute dyspnoea, circulatory failure or trauma, which are treated by air rescue physicians will be included in this study. Duration of ultrasound performance as well as altered treatment strategies will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patients suffering from acute dyspnoea, circulatory failure or trauma will be included.

Patients with acute dyspnoea will be included, if they show at least one of the two following signs of respiratory failure:

* Respiratory rate > 20 breaths per minute
* Peripheral oxygen saturation without oxygen supplementation < 90%

Patients with acute circulatory failure will be included, if they show at least one of the following signs:

* Hypotension (systolic blood pressure <90mmHg)
* Altered tissue perfusion (cold, clammy, mottling skin or altered mental status)

Trauma patients will be included, if at least one cause is suspected:

* Intraabdominal fluid
* Intrathoracic free fluid
* Pneumothorax

Exclusion Criteria:

* age under 18
* if POCUS will lead to a delay of live-saving treatment or transportation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 critically ill patients with acute dyspnoea, circulatory failure or trauma, will be included in this study. In 50 patients POCUS with tele-supervision and in 50 patients POCUS without tele-supervision will be performed. Tele-supervision is available in 50% of the time. Allocation to one of the two groups depends on the availability of tele-supervision.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of prehospital ultrasound between POCUS with or without tele-supervision | through study completion, an average of 1 year
  duration of prehospital ultrasound between POCUS with tele-supervision and POCUS without tele-supervision in critically ill patients (acute dyspnoea, circulatory failure, trauma).

SECONDARY OUTCOMES:
Alteration of treatent strategies | through study completion, an average of 1 year
  Investigating the impact of POCUS with tele-supervision in comparison to POCUS without tele-supervision on alteration of treatment strategies.

OTHER OUTCOMES:
Accuracy of suspected diagnosis in comparison to clinical findings | through study completion, an average of 1 year
  Investigating the impact of POCUS with tele-supervision in comparison to POCUS without tele-supervision on accuracy of suspected diagnosis in comparison to clinical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Department of Anaesthesia & General Intensive Care, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Anaesthesia & General Intensive Care, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided